CLINICAL TRIAL: NCT04419506
Title: A Randomised, Double-blind, Placebo-controlled Parallel Group Study in IPF Patients Over 12 Weeks Evaluating Efficacy, Safety and Tolerability of BI 1015550 Taken Orally
Brief Title: A Study to Test How Taking BI 1015550 for 12 Weeks Affects Lung Function in People With Idiopathic Pulmonary Fibrosis (IPF)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1305-0013; 2019-004167-45 (EudraCT Number)
Record Dates: First submitted 2020-06-04; First posted 2020-06-05 (Actual); Results first posted 2022-11-01 (Actual); Last update posted 2022-11-01 (Actual); Status verified 2022-10

CONDITIONS: Idiopathic Pulmonary Fibrosis
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis | interventions — BI 1015550

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Placebo, Antifibrotics at baseline (Placebo Comparator): Idiopathic pulmonary fibrosis (IPF) patients on stable antifibrotic treatment with nintedanib or pirfenidone at baseline were administered placebo matching BI 1015550 taken orally as film-coated tablets (matching the respective BI 1015550 tablets) twice daily, in the morning and in the evening for 12 weeks. During the 12-weeks of administration of BI 1015550 patients stayed on their stable background therapy of nintedanib or prifenidone.
  Interventions: Drug: Placebo
- BI 1015550, Antifibrotics at baseline (Experimental): Idiopathic pulmonary fibrosis (IPF) patients on stable antifibrotic treatment with nintedanib or pirfenidone at baseline were administered 18 milligram (mg) BI 1015550 taken orally as film-coated tablets (1x 6mg tablet, 1x 12 mg tablet) twice daily (36 mg daily), in the morning and in the evening for 12 weeks. During the 12-weeks of administration of BI 1015550 patients stayed on their stable background therapy of nintedanib or prifenidone.
  Interventions: Drug: BI 1015550
- Placebo, Non-antifibrotics at baseline (Placebo Comparator): Idiopathic pulmonary fibrosis (IPF) patients not on stable antifibrotic treatment at baseline were administered placebo matching BI 1015550 taken orally as film-coated tablets (matching the respective BI 1015550 tablets) twice daily, in the morning and in the evening for 12 weeks.
  Interventions: Drug: Placebo
- BI 1015550, Non-antifibrotics at baseline (Experimental): Idiopathic pulmonary fibrosis (IPF) patients not on stable antifibrotic treatment at baseline were administered 18 milligram (mg) BI 1015550 taken orally as film-coated tablets (1x 6mg tablet, 1x 12 mg tablet) twice daily (36 mg daily), in the morning and in the evening for 12 weeks.
  Interventions: Drug: BI 1015550

INTERVENTIONS:
Drug: BI 1015550 — 18 milligram (mg) BI 1015550 taken orally as film-coated tablets (1x 6mg tablet, 1x 12 mg tablet) twice daily (36 mg daily), in the morning and in the evening for 12 weeks.
  Arms: BI 1015550, Antifibrotics at baseline; BI 1015550, Non-antifibrotics at baseline
Drug: Placebo — placebo matching BI 1015550 taken orally as film-coated tablets (matching the respective BI 1015550 tablets) twice daily, in the morning and in the evening for 12 weeks.
  Arms: Placebo, Antifibrotics at baseline; Placebo, Non-antifibrotics at baseline

SUMMARY:
This study is open to adults with idiopathic pulmonary fibrosis (IPF) who are at least 40 years old. People taking standard medicines for IPF, including antifibrotic medicines, can continue taking them throughout the study.

The purpose of the study is to find out whether a medicine called BI 1015550 can slow down the worsening of lung function. Participants are in the study for about 4 months. During this time, they visit the study site about 7 times. At the beginning, they visit the study site every 2 weeks.

After 1 month of treatment, they visit the study site every 4 weeks.

The participants are put into 2 groups by chance. 1 group gets BI 1015550. The other group gets placebo. Placebo tablets look like BI 1015550 tablets but contain no medicine. The participants take BI 1015550 or placebo tablets twice a day.

The participants have lung function tests at study visits. The results of the lung function tests are compared between the BI 1015550 group and the placebo group. The doctors also regularly check the general health of the participants.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged ≥40 years when signing the informed consent.
2. Diagnosis:

   1. IPF based on 2018 ATS/ERS/JRS/ALAT Guideline as confirmed by the investigator based on chest High Resolution Computed Tomography Scan (HRCT) scan taken within 12 months of Visit 1 and if available surgical lung biopsy.

      and
   2. Usual interstitial pneumonia (UIP) or probable UIP HRCT pattern consistent with the clinical diagnosis of IPF, as confirmed by central review prior to Visit 2*

      * if indeterminate HRCT finding IPF may be confirmed locally by (historical) biopsy
3. Stable for at least 8 weeks prior to Visit 1. Patients have to be either :

   * not on therapy with nintedanib or pirfenidone for at least 8 weeks prior to Visit 1 (combination of nintedanib plus pirfenidone not allowed), or
   * on stable* therapy with nintedanib or pirfenidone for at least 8 weeks prior to Visit 1 and planning to stay stable on this background therapy after randomisation.

   [*stable therapy is defined as the individually and general tolerated regimen of either pirfenidone or nintedanib]
4. Forced Vital Capacity (FVC) ≥45% of predicted normal at Visit 1
5. Diffusion capacity of the lung for carbon monoxide (DLCO) (corrected for haemoglobin [Hb] [Visit 1]) ≥ 25% to < 80% of predicted normal at Visit 1.
6. Signed and dated written informed consent in accordance with ICH-GCP and local legislation prior to admission to the trial.

Exclusion Criteria:

1. Relevant airways obstruction (pre-bronchodilator Forced Expiratory Volume in one second (FEV1)/Forced Vital Capacity (FVC) < 0.7) at Visit 1.
2. In the opinion of the Investigator, other clinically significant pulmonary abnormalities.
3. Acute IPF exacerbation within 4 months prior to screening and/or during the screening period (investigator-determined).
4. Lower respiratory tract infection requiring antibiotics within 4 weeks prior to Visit 1 and/or during the screening period.
5. Major surgery (major according to the investigator's assessment) performed within 3 months prior to Visit 1 or planned during the course of the trial. (Being on a transplant list is allowed).
6. Any documented active or suspected malignancy or history of malignancy within 5 years prior to Visit 1, except appropriately treated basal cell carcinoma of the skin, "under surveillance" prostate cancer or in situ carcinoma of uterine cervix.
7. Evidence of active infection (chronic or acute) based on clinical exam or laboratory findings at Visit 1 or at Visit 2.
8. Any suicidal behaviour in the past 2 years (i.e. actual attempt, interrupted attempt, aborted attempt, or preparatory acts or behavior).
9. The patient has a confirmed infection with SARS-CoV-2 within the 4 weeks prior to Visit 1 and/or during the screening period.

Further exclusion criteria apply.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 147 (Actual)
Dates: Start 2020-07-28 (Actual); Primary Completion 2021-10-06 (Actual); Study Completion 2021-10-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (75):
- United States (11):
  - St. Francis Medical Institute, Clearwater, Florida
  - University of Florida, Gainesville, Florida
  - University of Kansas Medical Center, Kansas City, Kansas
  - Mayo Clinic, Rochester, Rochester, Minnesota
  - The Lung Research Center, LLC, Chesterfield, Missouri
  - Creighton University, Omaha, Nebraska
  - Southeastern Research Center, Winston-Salem, North Carolina
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - Temple University Hospital, Philadelphia, Pennsylvania
  - Diagnostics Research Group, San Antonio, Texas
  - University of Utah Health Sciences Center, Salt Lake City, Utah
- Centro de Investigaciones Metabólicas (CINME), C.a.b.a, Argentina
- The Alfred Hospital, Melbourne, Victoria, Australia
- LKH-Univ. Hospital Graz, Graz, Austria
- Canada (5):
  - St. Paul's Hospital, Vancouver, British Columbia
  - Dr. Georges-L.-Dumont University Hospital Centre, Moncton, New Brunswick
  - Queen's University, Kingston, Ontario
  - Dr. Syed Anees Medicine Professional Corporation, Windsor, Ontario
  - Centre Hospitalier de l'Universite de Montreal (CHUM), Montreal, Quebec
- Chile (2):
  - Instituto Nacional del Tórax, Providencia, Santiago de Chile
  - Centro de Investigación del Maule, Talca
- China (5):
  - Peking Union Medical College Hospital, Beijing
  - The Second Hospital of Jilin University, Changchun
  - West China Hospital, Chengdu
  - Zhongshan Hospital Fudan University, Shanghai
  - Shanghai Pulmonary Hospital, Shanghai
- Czechia (2):
  - University Hospital Na Bulovce, Prague, Prague
  - University Thomayer's Hospital, Praha 4 - Krc
- Denmark (3):
  - Aarhus University Hospital, Aarhus N
  - Herlev and Gentofte Hospital, Hellerup
  - Odense University Hospital, Odense C
- Finland (5):
  - HYKS Keuhkosairauksien tutkimusyksikkö, Helsinki
  - KYS, Keuhkosairauksien, Kuopio
  - Oulun yliopistollinen keskussairaala, Oulu
  - Tampere University Hospital, Tampere
  - TYKS, Turku
- Germany (5):
  - Fachkrankenhaus Coswig GmbH, Coswig
  - Ruhrlandklinik, Westdeutsches Lungenzentrum am Universitätsklinikum Essen gGmbH, Essen
  - Thoraxklinik-Heidelberg gGmbH am Universitätsklinikum Heidelberg, Heidelberg
  - Lungenfachklinik Immenhausen, Immenhausen
  - Universitätsklinikum Münster, Münster
- Greece (3):
  - Athens Medical Center, Athens
  - University General Hospital of Heraklion, Crete
  - Univ. Gen. Hosp. of Patras, Pátrai
- Semmelweis University, Budapest, Hungary
- Italy (4):
  - Ospedale Colonnello D Avanzo, Foggia
  - Azienda Ospedaliera Universitaria di Padova, Padua
  - Poli Univ A. Gemelli, Roma
  - A.O.U. Senese Policlinico Santa Maria alle Scotte, Siena
- Japan (6):
  - Tosei General Hospital, Aichi, Seto
  - National Hospital Organization Kyushu Medical Center, Fukuoka, Fukuoka
  - Kanagawa Cardiovascular and Respiratory Center, Kanagawa, Yokohama
  - National Hospital Organization Kinki-Chuo Chest Medical Center, Osaka, Sakai
  - Hamamatsu University Hospital, Shizuoka, Hamamatsu
  - Center Hospital of the National Center for Global Health and Medicine, Tokyo, Shinjuku-ku
- Netherlands (3):
  - Zuyderland Medisch Centrum, Heerlen
  - St. Antonius ziekenhuis, locatie Nieuwegein, Nieuwegein
  - Erasmus Medisch Centrum, Rotterdam
- University Clinical Center, Gdansk, Gdansk, Poland
- Russia (3):
  - Federal state budgetary scientific institution "Research Institute of occupational medicine named after academician N. F. Izmerov, Moscow
  - Moscow 1st State Med.Univ.n.a.I.M.Sechenov, Moscow
  - Emergency Clinical Hospital n. a. N. V. Solovyev, Yaroslavl, Yaroslavl
- South Korea (3):
  - The Catholic University of Korea, Bucheon St.Mary's Hospital, Bucheon-si
  - Seoul National University Hospital, Seoul
  - Asan Medical Center, Seoul
- Spain (6):
  - Policlínica Barcelona, Barcelona
  - Hospital Clínic de Barcelona, Barcelona
  - Hospital de Bellvitge, L'Hospitalet de Llobregat
  - Hospital La Princesa, Madrid
  - Hospital Central de Asturias, Oviedo
  - Hospital Son Espases, Palma de Mallorca
- Ukraine (2):
  - Dnyepropyetrovsk Medical Academy, Clinical Hospital No. 6, Dnyepropyetrovsk
  - Instit.Phthisiology&Pulmon.na Yanovskiy,Non-Specif.Lung,Kyiv, Kyiv
- United Kingdom (2):
  - Southmead Hospital, Bristol
  - Royal Brompton Hospital, London

IPD SHARING:
Plan to Share IPD: Yes
After the study is completed and the primary manuscript is accepted for publishing, researchers can use this following link https://www.mystudywindow.com/msw/datasharing to request access to the clinical study documents regarding this study, and upon a signed "Document Sharing Agreement".
  Also, Researchers can use the following link https://www.mystudywindow.com/msw/datasharing to find information in order to request access to the clinical study data, for this and other listed studies, after the submission of a research proposal and according to the terms outlined in the website.
  The data shared are the raw clinical study data sets.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: After all regulatory activities are completed in the US and EU for the product and indication, and after the primary manuscript has been accepted for publication.
Access Criteria: For study documents - upon signing of a 'Document Sharing Agreement'. For study data - 1. after the submission and approval of the research proposal (checks will be performed by both the independent review panel and the sponsor, including checking that the planned analysis does not compete with sponsor's publication plan); 2. and upon signing of a 'Data Sharing Agreement'.
URL: https://www.mystudywindow.com/msw/datasharing

REFERENCES:
- [Derived] Richeldi L, Azuma A, Cottin V, Hesslinger C, Stowasser S, Valenzuela C, Wijsenbeek MS, Zoz DF, Voss F, Maher TM; 1305-0013 Trial Investigators. Trial of a Preferential Phosphodiesterase 4B Inhibitor for Idiopathic Pulmonary Fibrosis. N Engl J Med. 2022 Jun 9;386(23):2178-2187. doi: 10.1056/NEJMoa2201737. Epub 2022 May 15. PMID 35569036
- See also: Related Info — http://mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a trial with a randomised, placebo-controlled, double-blind, parallel-group design over 12 weeks, including a screening period of up to 44 days, a 12-week treatment period, and a 1-week follow-up period in patients with idiopathic pulmonary fibrosis (IPF) stratified by baseline antifibrotic treatment (Non-AF stratum: patients not on antifibrotic treatment at baseline; AF stratum: stable antifibrotic treatment with nintedanib or pirfenidone at baseline).
Pre-assignment Details: All subjects were screened for eligibility prior to participation in the trial. Subjects attended a specialist site which ensured that they (the subjects) strictly met all inclusion and none of the exclusion criteria. Subjects were not to be allocated to a treatment group if any of the entry criteria were violated.
Groups:
- Placebo - Antifibrotics at Baseline: Idiopathic pulmonary fibrosis (IPF) patients on antifibrotic treatment with nintedanib or pirfenidone at baseline were administered placebo matching BI 1015550 taken orally as film-coated tablets (matching the respective BI 1015550 tablets) twice daily, in the morning and in the evening for 12 weeks. During the 12-weeks of administration of BI 1015550 patients stayed on their background therapy of nintedanib or prifenidone.
- BI 1015550 - Antifibrotics at Baseline: Idiopathic pulmonary fibrosis (IPF) patients on antifibrotic treatment with nintedanib or pirfenidone at baseline were administered 18 milligram (mg) BI 1015550 taken orally as film-coated tablets (1x 6mg tablet, 1x 12 mg tablet) twice daily (36 mg daily), in the morning and in the evening for 12 weeks. During the 12-weeks of administration of BI 1015550 patients stayed on their background therapy of nintedanib or prifenidone.
- Placebo - Non-antifibrotics at Baseline: Idiopathic pulmonary fibrosis (IPF) patients not on antifibrotic treatment at baseline were administered placebo matching BI 1015550 taken orally as film-coated tablets (matching the respective BI 1015550 tablets) twice daily, in the morning and in the evening for 12 weeks. Patients were not expected to start antifibrotic treatment during the 12 weeks of placebo treatment.
- BI 1015550 - Non-antifibrotics at Baseline: Idiopathic pulmonary fibrosis (IPF) patients not on antifibrotic treatment at baseline were administered 18 milligram (mg) BI 1015550 taken orally as film-coated tablets (1x 6mg tablet, 1x 12 mg tablet) twice daily (36 mg daily), in the morning and in the evening for 12 weeks. Patients were not expected to start antifibrotic treatment during the 12 weeks of BI 1015550 treatment.
Period: Overall Study
Arm/Group | Placebo - Antifibrotics at Baseline | BI 1015550 - Antifibrotics at Baseline | Placebo - Non-antifibrotics at Baseline | BI 1015550 - Non-antifibrotics at Baseline
Started | 25 | 49 | 25 | 48
Completed (Completion of trial medication) | 25 | 39 | 25 | 43
Not Completed | 0 | 10 | 0 | 5
Not completed — Adverse Event | 0 | 10 | 0 | 3
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1
Not completed — poor-compliance | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Treated Set (TS): all patients who received at least one dose of trial drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo - Antifibrotics at Baseline | BI 1015550 - Antifibrotics at Baseline | Placebo - Non-antifibrotics at Baseline | BI 1015550 - Non-antifibrotics at Baseline | Total
Number analyzed (Participants) | 25 | 49 | 25 | 48 | 147
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.5 (10.7) | 69.3 (6.6) | 71.8 (9.3) | 69.9 (8.3) | 69.6 (8.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 5 | 8 | 14 | 34
  Male | 18 | 44 | 17 | 34 | 113
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 3 | 4 | 5 | 13
  Not Hispanic or Latino | 24 | 46 | 21 | 43 | 134
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 4 | 12 | 4 | 12 | 32
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 21 | 37 | 21 | 36 | 115
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Forced vital capacity (FVC) [Mean (Standard Deviation); unit: Milliliter] — Forced vital capacity (FVC) at baseline. FVC is the total amount of air exhaled during a Forced expiratory volume (FEV) test. Population: Treated Set (TS): all patients who received at least one dose of trial drug.
  Milliliter | 2690.000 (889.985) | 2875.551 (752.818) | 2864.920 (1015.104) | 2782.938 (835.104) | 2811.946 (845.625)

OUTCOME MEASURES:

1. Primary Outcome: The Change From Baseline in Forced Vital Capacity (FVC) at 12 Weeks
Description: The change from baseline in Forced vital capacity (FVC) at 12 weeks. Data were analysed with a restricted maximum likelihood (REML)-based approach using a mixed model with repeated measures (MMRM). The analysis included the fixed, categorical effect of treatment at each visit, and the fixed, continuous effects of baseline FVC at each visit. Visit was treated as the repeated measure, with an unstructured covariance structure used to model the within-patient measurements.
Time Frame: Baseline (day 1) and week 12.
Population: Full Analysis Set (FAS): all patients who received at least one dose of trial drug and who had a baseline and at least one post-baseline measurement available for Forced Vital Capacity (FVC), Forced Expiratory Volume in one second (FEV1) or Diffusion Capacity of the Lung for Carbon Monoxide (DLCO).
Measure: Mean (95% Confidence Interval); unit: Milliliter
Arm/Group | Placebo - Antifibrotics at Baseline | BI 1015550 - Antifibrotics at Baseline | Placebo - Non-antifibrotics at Baseline | BI 1015550 - Non-antifibrotics at Baseline
Number analyzed (Participants) | 25 | 48 | 25 | 47
Milliliter | -77.70 [-124.87 to -30.53] | 2.72 [-33.46 to 38.89] | -95.62 [-157.13 to -34.10] | 6.10 [-39.67 to 51.88]
Statistical Analysis 1: Comparison: Placebo - Non-antifibrotics at Baseline vs BI 1015550 - Non-antifibrotics at Baseline; Adjusted means in the placebo group were combined with the meta-analytic predictive priors derived based on the clinical trials in the nintedanib clinical development program in IPF. In order to evaluate the treatment effects, the posterior distribution for the treatment difference of BI 1015550 versus placebo with respect to the primary endpoint was used. The median of the posterior distribution for the treatment difference (and 95% credible intervals) was calculated; Test type: Other; Posterior difference = 88.4, 95% CI 2-sided [29.5 to 154.2] — Difference calculated as BI 1015550 - Placebo
Statistical Analysis 2: Comparison: Placebo - Antifibrotics at Baseline vs BI 1015550 - Antifibrotics at Baseline; [analysis description as in outcome 1, analysis 1]; Test type: Other; Posterior difference = 62.4, 95% CI 2-sided [6.3 to 125.5] — Difference calculated as BI 1015550 - Placebo

2. Secondary Outcome: The Number of Patients With Treatment Emergent Adverse Event
Description: The number of patients with any adverse event during the on-treatment period.
Time Frame: From the start of treatment till the end of treatment + 7 days residual effect period, an average of 87.4 days.
Population: Treated Set (TS): all patients who received at least one dose of trial drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo - Antifibrotics at Baseline | BI 1015550 - Antifibrotics at Baseline | Placebo - Non-antifibrotics at Baseline | BI 1015550 - Non-antifibrotics at Baseline
Number analyzed (Participants) | 25 | 49 | 25 | 48
Participants | 5 | 18 | 5 | 9

ADVERSE EVENTS:
Time Frame: From the start of treatment till the end of treatment + 7 days residual effect period, an average of 87.4 days.
Description: Treated Set (TS): all patients who received at least one dose of trial drug.
Arm/Group | Placebo - Antifibrotics at Baseline | BI 1015550 - Antifibrotics at Baseline | Placebo - Non-antifibrotics at Baseline | BI 1015550 - Non-antifibrotics at Baseline
All-Cause Mortality (participants affected / at risk) | 0/25 | 1/49 | 0/25 | 1/48
Serious Adverse Events (participants affected / at risk) | 0/25 | 3/49 | 5/25 | 3/48
Other Adverse Events (participants affected / at risk) | 10/25 | 24/49 | 5/25 | 18/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo - Antifibrotics at Baseline (N=25) | BI 1015550 - Antifibrotics at Baseline (N=49) | Placebo - Non-antifibrotics at Baseline (N=25) | BI 1015550 - Non-antifibrotics at Baseline (N=48)
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 0 | 1
Condition aggravated (General disorders) | 0 | 2 | 0 | 0
COVID-19 pneumonia (Infections and infestations) | 0 | 0 | 0 | 1
Urosepsis (Infections and infestations) | 0 | 0 | 1 | 0
Wound infection (Infections and infestations) | 0 | 0 | 1 | 0
Diabetic metabolic decompensation (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Peripheral nerve paresis (Nervous system disorders) | 0 | 1 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Dermatitis exfoliative (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Vasculitis (Vascular disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo - Antifibrotics at Baseline (N=25) | BI 1015550 - Antifibrotics at Baseline (N=49) | Placebo - Non-antifibrotics at Baseline (N=25) | BI 1015550 - Non-antifibrotics at Baseline (N=48)
Constipation (Gastrointestinal disorders) | 2 | 1 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 4 | 15 | 2 | 8
Dyspepsia (Gastrointestinal disorders) | 1 | 2 | 0 | 3
Flatulence (Gastrointestinal disorders) | 1 | 2 | 1 | 3
Nausea (Gastrointestinal disorders) | 0 | 1 | 2 | 2
Asthenia (General disorders) | 0 | 1 | 0 | 3
Fatigue (General disorders) | 3 | 1 | 1 | 2
Nasopharyngitis (Infections and infestations) | 0 | 4 | 0 | 0
Headache (Nervous system disorders) | 1 | 3 | 0 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 4 | 1 | 3
Rash (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2020-09-09): https://cdn.clinicaltrials.gov/large-docs/06/NCT04419506/Prot_000.pdf
  • Statistical Analysis Plan (2021-10-08): https://cdn.clinicaltrials.gov/large-docs/06/NCT04419506/SAP_001.pdf